CLINICAL TRIAL: NCT01534416
Title: Use of Paracervical Block in Laparoscopic Gynecologic Surgery: A Randomized Controlled Trial
Brief Title: Effect of Paracervical Block on Post Operative Pain in Laparoscopic Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GCO 11-0021; HS# 11-00013
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain; Paracervical Block; Laparoscopic Gynecologic Surgery
Keywords: Paracervical Block; Laparoscopic Surgery; Postoperative Pain; Bupivacaine; Hysterectomy; Myomectomy; Randomized Trial
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Experimental): Subjects receive paracervical block with bupivacaine-epinephrine
  Interventions: Drug: Bupivacaine
- Saline (Placebo Comparator): Subjects receive paracervical injection of normal saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Bupivacaine — Subjects are injected paracervically with 10 ml of 0.5% bupivacaine with 1:200000 units epinephrine prior to surgical incision.
  Other Names: Marcaine
  Arms: Bupivacaine
Drug: Normal Saline — Subjects are injected paracervically with 10 ml of normal saline prior to surgical incision.
  Other Names: Saline
  Arms: Saline

SUMMARY:
The purpose of this study is to determine the effectiveness of placing numbing medication around the cervix prior to performing laparoscopic gynecologic surgery in decreasing pain after surgery. The study focuses on laparoscopic hysterectomies and robotic-assisted myomectomies. It will assess whether patients who receive the medication experience less pain and require less pain medication post operatively and if it helps reduce the number of patients who require hospitalization for pain control following surgery.

DETAILED DESCRIPTION:
A variety of traditionally open surgical procedures have recently become minimally invasive through the use of laparoscopic technology. Gynecologic surgeries are no exception. However, some gynecologic laparoscopic procedures are associated with significant post-operative pain, necessitating prolonged hospitalization, use of post-operative opioids, and in some cases, the development of chronic post-operative pain. Prolonged hospitalization and use of opioids pose important patient safety concerns, such as increased risk of hospital borne illnesses and medication errors; in addition, opioids may cause respiratory depression and addiction. Given the rising cost of health care there is also an economic incentive to eliminate the need for hospital admission due to post-operative pain.

Preemptive analgesia involves nerve blockade or administration of pain medication systemically prior to incision to reduce post-procedure pain. Paracervical blockade is a form of preemptive analgesia. Paracervical blocks have been demonstrated to be safe and effective for obstetrical procedures in reducing post-operative pain since the 1970s. Recently they have also been shown to be efficacious for reducing post-operative pain in vaginal hysterectomy (Long et al, Int Urogynecol J (2009) 20:5-10).

For the present investigation, we intend to study the effectiveness of paracervical blockade for laparoscopic and robotic-assisted laparoscopic gynecological surgery. We hypothesize that paracervical blockade prior to surgical incision will lessen levels of post-operative pain, reduce use of opioids, and decrease the number of patients requiring hospitalization for pain control. We also hypothesize that the effects may be longer lasting than the immediate post-operative period and may decrease the amount of time to return to normal activity after surgery.

Using anecdotal evidence from the primary investigator, Dr. Ascher-Walsh the rate of hospitalization for laparoscopic hysterectomy (laparoscopic-assisted vaginal hysterectomy, total laparoscopic hysterectomy, laparoscopic assisted supracervical hysterectomy) is approximately 67%. In this study, we wish to decrease hospitalization with the paracervical block by 50%, thus obtaining an overall post-operative hospitalization rate of 33%. For robotic-assisted laparoscopic myomectomy, the rate of hospitalization is 50%. We wish to decrease this by 50% as well. Overall we are aiming to achieve a rate of 30% for post-operative hospitalization for pain control for laparoscopic hysterectomies and robotic myomectomies combined.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 or older
* Scheduled for robotic-assisted laparoscopic myomectomy or laparoscopic hysterectomy, including total and supracervical hysterectomy, laparoscopic-assisted vaginal hysterectomy
* Surgery being performed for benign disease

Exclusion Criteria:

* Male
* Women under 18 years old
* Pregnancy
* Suspected or known malignant disease
* Immunocompromised

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Long JB, Eiland RJ, Hentz JG, Mergens PA, Magtibay PM, Kho RM, Magrina JF, Cornella JL. Randomized trial of preemptive local analgesia in vaginal surgery. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jan;20(1):5-10. doi: 10.1007/s00192-008-0716-6. Epub 2008 Oct 2. PMID 18830553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing laparoscopic surgery for benign indications were enrolled between 2011 and 2013
Groups:
- Bupivacaine: Subjects received a 20mL paracervical injection of 0.25% bupivacaine with 1:200000 units epinephrine prior to surgical incision.
- Saline: Subjects injected paracervically with 10 ml of normal saline prior to surgical incision.
Period: Overall Study
Arm/Group | Bupivacaine | Saline
Started | 68 | 64
Completed | 68 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Saline | Total
Number analyzed (Participants) | 68 | 64 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.2) | 47.8 (9.3) | 48.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 64 | 132
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 36 | 28 | 64
  Black | 12 | 20 | 32
  Hispanic | 13 | 10 | 23
  Asian | 4 | 3 | 7
  Other | 2 | 2 | 4
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (5.7) | 29.1 (6.9) | 28.1 (6.4)
Parity [Count of Participants; unit: Participants]
  0 | 21 | 38 | 59
  1 | 10 | 10 | 20
  2 | 22 | 19 | 41
  ≥3 | 15 | 11 | 26
Surgical Indication [Count of Participants; unit: Participants]
  Fibroids | 7 | 9 | 16
  Bleeding | 2 | 1 | 3
  Prolapse | 14 | 8 | 22
  Pain | 4 | 1 | 5
  Other | 0 | 3 | 3
  Fibroids & bleeding | 19 | 14 | 33
  Fibroids, bleeding & pain | 18 | 23 | 41
  Bleeding & pain | 4 | 5 | 9
Uterine Size [Mean (Standard Deviation); unit: weeks] | 13.7 (5.5) | 14.2 (4.6) | 14.0 (5.1)
Preoperative Hematocrit [Mean (Standard Deviation); unit: % of cells] | 36.8 (4.0) | 36.6 (4.2) | 36.7 (4.1)
Admission Planned [Number; unit: admissions] — planned overnight admission for non-medical reasons
  admissions | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital Admission for Postoperative Pain Control
Description: Unplanned hospital admissions and the hospital admissions at the request of the patients for pain management
Time Frame: Four hours after conclusion of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Saline
Number analyzed (Participants) | 68 | 64
Participants
  Unplanned admission | 23 | 17
  Unplanned admission for pain | 10 | 11

2. Secondary Outcome: Postoperative Pain Score
Description: Postoperative pain levels assessed using the visual analogue pain scale. This scale pairs faces with numbers 1-10, with 1 being no pain and 10 being extreme pain. In the PACU pain assessed using this scale by the nursing staff.
Time Frame: 1and 2 hour postoperatively
Population: This doesn't include hospitalization for reasons other than pain management.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bupivacaine: Subjects received a 20mL paracervical injection of 0.25% bupivacaine with 1:200000 units epinephrine prior to surgical incision and admitted for pain management.
  Participants who requested admission specifically for pain management.
- Bupivacaine Discharged: Subjects who received bupivacaine and epinephrine and discharged home after surgery. Participants in the Bupivacaine arm who were not admitted.
- Saline Group: Subjects injected paracervically with 10 ml of normal saline prior to surgical incision who were admitted for pain management. participants in the Saline arm who requested admission specifically for pain management.
- Saline Discharged Participants: Subjects who received saline and discharged after surgery. Participants in the Saline arm who were discharged after procedure and not admitted.
Arm/Group | Bupivacaine | Bupivacaine Discharged | Saline Group | Saline Discharged Participants
Number analyzed (Participants) | 10 | 40 | 11 | 46
units on a scale
  1 hour postoperative | 4.7 (2.9) | 3.9 (2.2) | 5.1 (2.0) | 4.5 (2.4)
  2 hours postoperative | 4.3 (2.5) | 2.7 (1.8) | 4.5 (2.4) | 3.8 (2.3)

3. Secondary Outcome: Postoperative Pain Score
Description: Postoperative pain levels assessed using the visual analogue pain scale. This scale pairs faces with numbers 1-10, with 1 being no pain and 10 being extreme pain. In the PACU pain assessed using this scale by the nursing staff. On postoperative days 1 and 2 the subjects self-reported their pain level.
Time Frame: 1, 2, 4 hour postoperatively, Day 1 post operatively, Day 2 postoperative
Population: Only those subjects with pain analyzed
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bupivacaine: Subjects received a 20mL paracervical injection of 0.25% bupivacaine with 1:200000 units epinephrine prior to surgical incision and admitted for pain management
- Saline Group: Subjects injected paracervically with 10 ml of normal saline prior to surgical incision who were admitted for pain management
Arm/Group | Bupivacaine | Saline Group
Number analyzed (Participants) | 64 | 59
units on a scale
  1 hour postoperative | 4.30 (2.55) | 4.69 (2.29)
  2 hours postoperative | 3.37 (2.19) | 4.01 (2.32)
  4 hours postoperative | 3.83 (2.57) | 4.35 (2.43)
  Day 1 postoperative | 3.80 (2.53) | 4.35 (2.14)
  Day 2 postoperative | 3.16 (2.34) | 3.37 (2.39)

4. Secondary Outcome: Postoperative Day Pain Medication Use
Description: Numbers of Patients Using Pain Medication on Postoperative Days 1-10. The subjects recorded at home the type and amount of pain medication they use for 10 days postoperatively.
Time Frame: Postoperative days 0-10
Population: missing data from 5 participants in Bupivacaine Arm and 4 in Saline Arm
Measure: Number; unit: participants
Groups:
- Bupivacaine OTC Analgesics Use: OTC - over-the-counter
Arm/Group | Bupivacaine Narcotics Use | Saline Narcotics Use | Bupivacaine OTC Analgesics Use | Saline OTC Analgesics Use
Number analyzed (Participants) | 63 | 60 | 63 | 60
participants
  Postoperative Day 1 | 52 | 52 | 17 | 10
  Postoperative Day 2 | 43 | 39 | 24 | 18
  Postoperative Day 3 | 28 | 33 | 29 | 22
  Postoperative Day 4 | 19 | 26 | 28 | 26
  Postoperative Day 5 | 13 | 15 | 19 | 28
  Postoperative Day 6 | 12 | 13 | 15 | 24
  Postoperative Day 7 | 5 | 11 | 16 | 16
  Postoperative Day 8 | 3 | 10 | 12 | 12
  Postoperative Day 9 | 2 | 6 | 9 | 11
  Postoperative Day 10 | 3 | 7 | 9 | 10

ADVERSE EVENTS:
Time Frame: Complications were noted up to 6 weeks after surgery using the Clavien-Dindo Classification system.
Description: Grade I Any deviation from normal postoperative course without need for pharmacological treatment or surgical, endoscopic, & radiological interventions II Require pharmacological treatment with drug other than such allowed for Grade I complications III Require surgical, endoscopic or radiological intervention IIIa Intervention not under general anaesthesia IIIb Intervention under general anaesthesia IV Life-threatening complication IVa Single organ IVb Multiorgan V Death
Arm/Group | Bupivacaine | Saline
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/68 | 0/64
Other Adverse Events (participants affected / at risk) | 17/68 | 16/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine (N=68) | Saline (N=64)
Stress Incontinence (Renal and urinary disorders) | 1 | 0 — Stress incontinence requiring a midurethral sling
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bupivacaine (N=68) | Saline (N=64)
Urinary Tract Infection (Renal and urinary disorders) | 0 | 3
Incisional Infection (Injury, poisoning and procedural complications) | 4 | 4
Urinary Retention (Renal and urinary disorders) | 6 | 6
Small Bowel Mesenteric Hematoma (Injury, poisoning and procedural complications) | 0 | 1 — a small bowel mesenteric hematoma caused by Veress needle injury that did not require surgical management
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 — skin laceration from the morcellator
Cervical infection (Reproductive system and breast disorders) | 2 | 1
Retropubic hematoma (Injury, poisoning and procedural complications) | 1 | 1
Bladder performation (Injury, poisoning and procedural complications) | 1 | 0 — bladder perforation during a concomitant retropubic midurethral sling procedure
Seizure (General disorders) | 1 | 0 — unknown etiology
Emergency Room Visit (General disorders) | 1 | 0 — ER visit for nausea, vomiting, and headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes